CLINICAL TRIAL: NCT02871895
Title: Application of Biomarkers Change to Predict Outcome of Patients With Severe Sepsis
Brief Title: Application of Biomarkers Change to Predict Outcome of Patient With Severe Sepsis
Acronym: BCSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8B1063
Record Dates: First submitted 2015-09-01; First posted 2016-08-18 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS); Sepsis; Severe Sepsis; Septic Shock; Multiple Organ Failure
Keywords: sepsis; severe sepsis; septic shock; multiple organ failure
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum immunological biomarkers including cytokines, blood cell counts,and biochemistry profiles
Oversight: Data Monitoring Committee: No

SUMMARY:
In 2004, the Surviving Sepsis Campaign (SSC) introduced guidelines for the management of severe sepsis and septic shock, as well as strategies for bedside implementation. The treatment recommendations were organized in two bundles. In an international study, enrolling adult patients with severe sepsis admitted to these intensive care units, investigators found that while mortality from severe sepsis is high (44.5%), compliance with resuscitation and management bundles is generally poor in much of Asia. Investigators need to identify the patients at risk for high in-hospital mortality in order to take appropriate steps.

From their past studies, investigators found that sepsis involved inflammation and coagulation. The multiple organ involvement was associated with interaction of novel biomarkers such as cytokines. There is limited data regarding comparing and application of biomarkers of different characteristic on sepsis treatment. A simultaneous detection of multiple cytokines may provide significant prognostic information. For other biomarkers, promising observation data have been put forward, but their potential needs to be evaluated in large-scale, well-designed prospective intervention studies before clinical use can be recommended. Besides many clinical studies on biomarkers were confounded by its lack of standard bundle care for severe sepsis patient.

Here investigators performed a systematic study aimed at evaluating

1. the individual and combined diagnostic accuracy of biomarkers for predicting mortality;
2. whether trend change in biomarker level more useful for above prediction;
3. which biomarker or biomarker combination checked can predict patients at risk of evolving with severe organ dysfunctions.

DETAILED DESCRIPTION:
Variables will be tested for their association with the outcome using Pearson chi-square test for categorical data and Mann-Whitney U test for numerical data. Comparison the different groups will be conducted by using Mann-Whitney U test for numerical data and using Pearson chi-square test for categorical data. The time course of biomarker plasma levels will be assessed by analysis of variance. Multivariate analysis will be performed using a logistic regression model to estimate the odds ratio of organ failure and dying, along with the 95% confidence interval (CI). Forward and backward selection procedures will be used to iteratively select the variables potentially related to death.

Discrimination will be assessed using the area under the receiver operating characteristic curve to evaluate how well the model distinguished patients who lived from those who died and whether progression of organ dysfunction. A survival analysis will be performed using Kaplan-Meier curves and the log-rank test. Analyses will be completed and a two-tailed p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis
* Septic shock

Exclusion Criteria:

* Patients are < 18 yrs
* Patients are immunocompromised (treatment with corticosteroids >1 mg/kg equivalent prednisone)
* Bone marrow or organ transplant recipients,
* Leucopenia [white blood cells count< 109/L] or neutropenia [polymorphonuclear granulocyte count <0.5 109/L]
* Hematologic malignancy
* Acquired immune deficiency syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Kaohsiung Chang Gung Memorial Hospital. All adult patients presenting with sepsis or severe sepsis will be enrolled on admission to medical intensive units (total 34 beds). Sepsis and severe sepsis are defined as American College of Chest Physicians/Society of Critical Care Medicine consensus criteria for sepsis syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Development of immune dysfunction score to predict 28-day mortality of sepsis patients | baseline and 4 weeks, up to 24 weeks
  Several existing scoring systems developed for mortality prediction, such as APACHE II and Sequential Organ Failure Assessment score (SOFA score). However, none of these take immune dysfunction status into account. With a substantial degree of heterogeneity in the sepsis response ranging from cytokines storm to immunoparalysis, better patient stratification is needed. Investigators aimed to develop and validate a scoring system (minimum:0 to maximum:6 scores) that can determine patients' immune dysfunction status related to outcomes.

SECONDARY OUTCOMES:
Deteriorated dynamic acute kidney injury (AKI) stage associated with immune dysfunction and higher mortality in Septic Patients Admitted to Intensive Care Unit | baseline and 4 weeks, up to 24 weeks
  A series of inflammatory cytokines participated into the mechanism and associated with the severity and worsening of AKI. We assumed the dynamic change of the AKI containing even better predictive value rather than evaluating the AKI in a single time point. We categorized septic patients into 4 groups based on the variation of AKI stage. In addition to mortality comparison, we also made an investigation to the relationships of immune cytokines in those sepsis patients.
To determine whether delta pulse pressure at day 3 compared with day 1 affect survival outcomes in patients who were diagnosed sepsis and septic shock. | baseline and 4 weeks
  Pulse pressure is the difference between the systolic and diastolic blood pressures. It arises from the interaction of cardiac ejection and the properties of the arterial circulation. A wide pulse pressure is associated with increased cardiovascular mortality. However, a widened pulse pressure was suggested as a potential prognostic indicator of decreased mortality in patients with sepsis in a retrospective electronic medical record review. In clinical practice, pulse pressure variation can help predict fluid responsiveness in patients. Furthermore, we sought to determine whether stratification of septic patients according to the changes of pulse pressure (value of pulse pressure at day 3 minus value of pulse pressure at day 1) and status of whether still in need of vasopressor at day 3 could help predict survival. The host immune response to sepsis during progression may play an important role.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Feng Fang, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Neveu H, Kleinknecht D, Brivet F, Loirat P, Landais P. Prognostic factors in acute renal failure due to sepsis. Results of a prospective multicentre study. The French Study Group on Acute Renal Failure. Nephrol Dial Transplant. 1996 Feb;11(2):293-9. doi: 10.1093/oxfordjournals.ndt.a027256. PMID 8700363
- [Result] Vincent JL, Abraham E, Annane D, Bernard G, Rivers E, Van den Berghe G. Reducing mortality in sepsis: new directions. Crit Care. 2002 Dec;6 Suppl 3(Suppl 3):S1-18. doi: 10.1186/cc1860. Epub 2002 Dec 5. PMID 12720570
- [Result] Salluh JI, Bozza PT. Biomarkers of sepsis: lost in translation? Crit Care Med. 2008 Jul;36(7):2192-4. doi: 10.1097/CCM.0b013e31817c0cd8. No abstract available. PMID 18594226
- [Result] Shiramizo SC, Marra AR, Durao MS, Paes AT, Edmond MB, Pavao dos Santos OF. Decreasing mortality in severe sepsis and septic shock patients by implementing a sepsis bundle in a hospital setting. PLoS One. 2011;6(11):e26790. doi: 10.1371/journal.pone.0026790. Epub 2011 Nov 3. PMID 22073193
- [Result] Nguyen HB, Corbett SW, Steele R, Banta J, Clark RT, Hayes SR, Edwards J, Cho TW, Wittlake WA. Implementation of a bundle of quality indicators for the early management of severe sepsis and septic shock is associated with decreased mortality. Crit Care Med. 2007 Apr;35(4):1105-12. doi: 10.1097/01.CCM.0000259463.33848.3D. PMID 17334251
- [Result] Phua J, Koh Y, Du B, Tang YQ, Divatia JV, Tan CC, Gomersall CD, Faruq MO, Shrestha BR, Gia Binh N, Arabi YM, Salahuddin N, Wahyuprajitno B, Tu ML, Wahab AY, Hameed AA, Nishimura M, Procyshyn M, Chan YH; MOSAICS Study Group. Management of severe sepsis in patients admitted to Asian intensive care units: prospective cohort study. BMJ. 2011 Jun 13;342:d3245. doi: 10.1136/bmj.d3245. PMID 21669950
- [Result] Jones AE, Puskarich MA. Is lactate the "Holy Grail" of biomarkers for sepsis prognosis? Crit Care Med. 2009 May;37(5):1812-3. doi: 10.1097/CCM.0b013e3181a09487. No abstract available. PMID 19373056
- [Result] Schuetz P, Haubitz S, Mueller B. Do sepsis biomarkers in the emergency room allow transition from bundled sepsis care to personalized patient care? Curr Opin Crit Care. 2012 Aug;18(4):341-9. doi: 10.1097/MCC.0b013e328354b2c8. PMID 22610364
- [Result] Kwak SH, Wang XQ, He Q, Fang WF, Mitra S, Bdeir K, Ploplis VA, Xu Z, Idell S, Cines D, Abraham E. Plasminogen activator inhibitor-1 potentiates LPS-induced neutrophil activation through a JNK-mediated pathway. Thromb Haemost. 2006 May;95(5):829-35. PMID 16676075
- [Result] Wang XQ, Bdeir K, Yarovoi S, Cines DB, Fang W, Abraham E. Involvement of the urokinase kringle domain in lipopolysaccharide-induced acute lung injury. J Immunol. 2006 Oct 15;177(8):5550-7. doi: 10.4049/jimmunol.177.8.5550. PMID 17015742
- [Result] Hoke TS, Douglas IS, Klein CL, He Z, Fang W, Thurman JM, Tao Y, Dursun B, Voelkel NF, Edelstein CL, Faubel S. Acute renal failure after bilateral nephrectomy is associated with cytokine-mediated pulmonary injury. J Am Soc Nephrol. 2007 Jan;18(1):155-64. doi: 10.1681/ASN.2006050494. Epub 2006 Dec 13. PMID 17167117
- [Result] Lin MC, Leung SY, Fang WF, Chin CH, Chung KF. Down-regulation of insulin-like growth factor I (IGF-I) in the mouse diaphragm during sepsis. Chang Gung Med J. 2010 Sep-Oct;33(5):501-8. PMID 20979700